CLINICAL TRIAL: NCT06291792
Title: Efficiency Of Otago Exercise Program Applied By Telerehabilitation Method In Older Persons Individuals With A Fall Story
Brief Title: Otago Exercise Program Applied By Telerehabilitation
Acronym: OEPABT
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Sinop University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: FTR001
Record Dates: First submitted 2023-07-12; First posted 2024-03-04 (Actual); Last update posted 2024-03-04 (Actual); Status verified 2024-02

CONDITIONS: Older People--Abuse of; Falling; Balance; Distorted
Keywords: Fear of Falling; Balance; Older Persons; Telerehabilitation; Otago Exercise

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Telerehabilitation Otago Exercise Group (TOEG) (Experimental): The use of Otago Exercise Program in the home environment using the telerehabilitation method. Telerehabilitation was performed with video and audio interviews 3 times a week for 45 minutes.
  The study will take 12 weeks. An 8-week treatment protocol will be applied. 4 weeks after the treatment protocol, the last measurement will be made and the study will be terminated.
  Interventions: Other: telerehabilitation otago exercise program
- Face to face Otago Exercise Group (FOEG) (Experimental): Otago Exercise Program was applied in a face-to-face clinical setting. Interviews were held 3 times a week for 45 minutes.
  The study will take 12 weeks. An 8-week treatment protocol will be applied. 4 weeks after the treatment protocol, the last measurement will be made and the study will be terminated.
  Interventions: Other: face to face otago exercise program

INTERVENTIONS:
Other: telerehabilitation otago exercise program — telerehabilitation otago exercise program
  Arms: Telerehabilitation Otago Exercise Group (TOEG)
Other: face to face otago exercise program — face to face otago exercise program
  Arms: Face to face Otago Exercise Group (FOEG)

SUMMARY:
The aim of this study is to examine the effects of Otago Exercise Program (OEP) on pain, walking speed, lower extremity muscle strength, fear of falling, anxiety, quality of life and balance with the telerehabilitation method in individuals with a history of falling, which is frequently seen in elderly individuals due to aging.

45 people between the ages of 65 and 78 participated in the study. They were randomly divided into 3 groups as control, telerehabilitation otago exercise program (TOEG) and face-to-face otago exercise program (FOEG). 45 minutes of OEP was applied 3 times a week for 8 weeks. Pain, walking speed, lower extremity muscle strength, fear of falling, anxiety, quality of life, and balance were evaluated before the Otago Exercise Program, at the 4th week, at the 8th week, and 4 weeks after the end of the exercise program. Significance was evaluated at the p<0.05 level in the study.

DETAILED DESCRIPTION:
Those using a randomized controlled clinical trial model that includes assessment methods over four different time periods. Detailed information about the procedure to be applied was given to each participant who would participate in the study. After the information, mini mental state test was applied to the participants who signed the consent form. Gender, age, weight, height, number of falls in the last 1 year, body mass indexes were calculated and recorded, including demographic information of the participants who met the inclusion criteria. Participants were randomly divided into 3 groups. The groups are; telerehabilitation otago exercise program (TOEG) (n=15, 8 males, 7 females), face-to-face otago exercise program (FOEG) (n=15, 8 males, 7 females), Control Group (CG) (n=15) , 8 men, 7 women).

ELIGIBILITY:
Inclusion Criteria:

* Presence of the ability to walk without assistance
* Living independently at home
* Having a history of at least one fall in the last 12 months

Exclusion Criteria:

* Having a score below 24 on the Mini Mental State Test
* Using a walking aid
* Having a history of uncontrolled epileptic seizures
* Having a history of surgery within the last six months

Ages: 65 Years to 90 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2023-11-01 (Actual); Primary Completion 2024-03-01 (Estimated); Study Completion 2024-03-01 (Estimated)

PRIMARY OUTCOMES:
Numerical Pain Scale | within 10 minutes after intervention
  Numerical pain scale is used to classify pain from 1 to 10. 1 represents the lowest and 10 represents the highest pain value.
Walking Speed | within 10 minutes after intervention
  Walking Speed
lower extremity muscle strength | within 10 minutes after intervention
  lower extremity muscle strength measurement; It is used to determine the strength rate of lower extremity muscles. Muscles are classified from 0 to 5 according to the resistance applied against them and the counter force they show. While 0 indicates the lowest muscle strength, 5 indicates the highest muscle strength.
Fall effectiveness scale | within 10 minutes after intervention
  There are 10 questions asked to the participant that are relevant to daily life at home. Each of the questions is answered numerically with a score between 1 and 10. The sum of the answers gives the total result of the test. If the result is higher than 70 points, the individual's fear of falling is high. As the fear of falling increases, the score of the test increases.
Beck anxiety scale | within 10 minutes after intervention
  This scale asks about situations related to the person's body that are indicative of anxiety, such as sweating, shaking, fear, and discomfort in various areas. There are a total of 21 questions and 4 verbal answers that can be given to each question. Each verbal response has 4 different numerical scores between 0 and 3. At the end of the test, the numerical scores of the answers are added up. The total score gives the result of the test. If it is less than 21 points, the anxiety is low, between 22 and 35 points, the anxiety is moderate, and if it is 36 and above, it is said that there is severe anxiety.
Tinetti balance and walking test | within 10 minutes after intervention
  It examines balance and walking status in 2 categories. There are 9 balance questions, followed by 7 questions about walking. There are 16 questions in total. A simple standard chair, a timer and a distance of about 15 meters is sufficient. Each question has 3 answers and each answer has numerical values of 0, 1, 2. The total score is calculated by adding the total score of the balance questions and the total score of the walking questions.
  The maximum score that balance questions can receive is 26, and the maximum score that walking questions can receive is 9. Total test score can be maximum 35. If the total test score is less than 18, it indicates a high risk of falling, if it is between 19-24, it indicates a slight risk, and if it is 24 and above, it indicates a low risk of falling.
World Health Organization Quality of Life Scale: | within 10 minutes after intervention
  This scale, developed for scientific research and clinical studies on the elderly, consists of 24 questions. It aims to measure the quality of life of the elderly individual. Each question has 5 verbal answers and each verbal answer has a numerical value between 1 and 5. At the end of the test, the numerical values of all answers are summed. The total score gives the result of the test. As the score of the test increases, the quality of life of the elderly participant also increases.

CONTACTS AND LOCATIONS:
Overall Officials: SEFA HAKTAN HATIK, PhD, Study Chair — Sinop University
Locations (1):
- Bahçeşehir University research application center, Istanbul, Turkey (Türkiye)